CLINICAL TRIAL: NCT03139539
Title: Intraoperative Microbial Contamination, Its Prevention and Its Consequences for Outcomes Following Joint Replacement Surgery
Brief Title: Intraoperative Microbial Contamination
Acronym: ICON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Frederiksberg University Hospital (Other); Hillerod Hospital, Denmark (Other); Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Anne Brun Hesselvig, MD, Primary Investigator, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-15012754
Record Dates: First submitted 2017-04-27; First posted 2017-05-04 (Actual); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Periprosthetic Joint Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ioban (Active Comparator): In this arm patients will be operated using Ioban as incisional drape.
  Interventions: Device: Ioban
- Control (No Intervention): In this arm patients will be operated using no incisional drape.

INTERVENTIONS:
Device: Ioban
  Other Names: iodine impregnated incisional foil
  Arms: Ioban

SUMMARY:
This is a randomized, controlled study which aims to show whether iodine impregnated incisional foil (IobanTM) has a place in the prevention of prosthetic joint infection (PJI). 1200 patients will be included in this study and will be followed through out a ten year period.

Follow up will center on the function of the prosthetic knee, early and late infection rates and revision surgery due to aseptic loosening.

Our purpose is to gain insight in to the causes of post-operative infection in joint alloplasty surgery. Our hypothesis' are:

1. The patient's skin flora is the main source of intraoperative contamination,
2. Intraoperative contamination can be reduced by using IobanTM
3. Intraoperative contamination strongly predicts postoperative infection
4. Unsuccessful clinical outcomes of knee arthroplasty are caused by low-grade infections.

To our knowledge this is the first study with this large a sample size and as long a follow up.

Background PJI is a devastating complication with substantial morbidity and high socio economic costs. Revision surgery due to infection costs as much as six times more than the primary surgery and has a poorer outcome for the patient i.e. disability, pain or loss of function.

Methods and materials

The study has two main arms:

1. Intraoperative contamination
2. Postoperative infection

The first stage aims to document that patients with intraoperative contamination have a larger risk of developing postoperative infection and include a study of the effect of Ioban™.

The second stage are to include methods of PCR (polymerase chain reaction) and fluorescence microscopy, to demonstrate bacterial contamination and/or infection of any implants removed during the study period.

Perspectives This study will give us new insight in the causes of PJI and the correlation with contamination during surgery. If IobanTM is proved to prevent infection it is a simple way to prevent post-operative infection and can be implemented in any orthopedic department.

DETAILED DESCRIPTION:
Introduction Approximately 8,000 primary knee arthroplasty procedures are performed annually at Danish hospitals (1). Infection is a serious complication that occurs with a frequency of around 2 %.

A mean of hindering infection is the use of IobanTM, an incisional drape impregnated with iodine. This costs 69 DKK pr. sheet. A two-stage stage operation for infection costs 253,122 DKK. (2) Using IobanTM for 8000 knee operations costs 552,000 DKK. Besides high socio economic costs infections cause considerable morbidity and have severe consequences for the independent mobility of the patient (3-5).

As the estimated number of arthroplasty procedures continuously increase so will the number of infections (6), and prevention is therefore of high priority.

Aim

The inestigators' purpose is to gain insight in to the causes of post-operative infection in joint arthroplasty surgery. The investigators' hypothesis' are:

1. The patient's skin flora is the main source for intraoperative microbial contamination,
2. Intraoperative contamination can be reduced by using an iodine impregnated incisional drape,
3. Intraoperative contamination strongly predicts postoperative infection
4. Unsuccessful clinical outcomes of knee arthroplasty are caused by low-grade infections.

Perspectives If intraoperative contamination can be shown to be a strong predictor of postoperative infection, then contamination will be an obvious outcome parameter for studies of preventive measures for infection. Demonstration of a strongly predictive role of intraoperative contamination may allow new prophylactic strategies for preventing postoperative infection, and one will have to consider prolonged antibiotic prophylaxis or treatment for patients, where contamination has been demonstrated.

Results of the study will provide information that will shape future strategies for preventing, diagnosing and treating peri-prosthetic joint infections.

The risk of adverse outcome for the participants is largely outweighed by the probability of discovering an early infection following surgery. This project's findings will be of great value for future patients undergoing knee replacement surgery.

Background and theory Recent studies have shown that a considerable proportion of orthopedic procedures performed under supposedly sterile conditions are contaminated. Contamination of the surgical field is found using swabs during surgery. There are several possible sources of intraoperative contamination. An obvious source is the patient's skin flora. Under normal circumstances, these bacteria are considered harmless, but in the presence of biomaterials like prosthetic implants, they have a significant pathogenic potential (7). It is well recognized that these bacteria adhere to the surface of the implant, where they multiply and transform into a biofilm formation making them more resistant to antibiotics and host defense mechanisms (8, 9). As a result they are involved in the development of low-grade persistent infections, which today still represent a major diagnostic challenge.

Furthermore, it is suggested that an unknown proportion of implant loosening are caused by infections of low virulence that do not result in recognizable infection (10). In this respect, reported infection rates are probably underestimated.

Standard procedures have been developed to reduce skin contamination including the use of preoperative skin antiseptics. However, even with optimal skin preparation, total sterilization of the skin is not possible. Some microorganisms will remain in the deeper parts of the skin, such as the hair follicles, and appear at the skin surface during surgery, where they will potentially contaminate the surgical field (11). One strategy of preventing microbial re-colonization on the skin is the application of an iodine impregnated incision drape preoperatively. In theory, this drape provides continuous antimicrobial activity throughout the surgical procedure thereby reducing skin contamination.

There are only few studies on the efficacy of iodine impregnated drapes. Some studies show reduced contamination rate with or without impact on infection rate. Other studies, however, have not been able to support this observation (12-14). All of these studies have had an insufficient amount of patients included. Consequently, there are no conclusions for standardized practice regarding the use of iodine impregnated incisions drapes. To clarify their correlation with intraoperative contamination as well as their preventive effect on the development of peri-prosthetic infection, large clinical trials are needed.

Cost benefit analysis One sheet of IobanTM costs 69 DKK. A two stage operation with removal of implant, implantation of a spacer and subsequent removal of spacer and implantation of a secondary implant costs 253.122 DKK (2). The one year revision rate I 1.8 % and a total of 8298 knees operated. Assuming half of these revisions are due to infection and are operated on using a two stage technique 18.731.028 DKK could be saved every year. These numbers are solely covering hospital expenses and not physiotherapy or rehabilitation or any other costs related to the surgery.

Using IobanTM in all patients undergoing total knee joint replacement costs 572.532 DKK a year. If this can prevent half of the one year revisions rates a total of 18.2 mio DKK could be saved each year. There is reason to believe that the investigators' findings could be extrapolated to other orthopedic procedures were implants are used saving the hospital large amounts of money on revisions every year. Not to mention the amount that could be saved on sickness benefit.

Feasibility An unpublished pilot study, performed by this research group, of 86 primary arthroplasty procedures showed a 10.5 % frequency of intraoperative contamination. Two of nine intra-operatively contaminated patients developed infection post-operatively, whereas only one of the 77 non-contaminated patients developed post-operative infection. A randomized sub-study showed that the use of an iodine impregnated incisional drape resulted in no intra-operative contamination in 19 patients compared to 3 cases of contamination in 11 patients operated without the use of an incisional drape.

400 patients are already included in this study and have been operated and have had samples taken. Preliminary results show a contamination rate of 5 %.

Samples will be collected at Orthopedic Departments at Herlev og Gentofte Hospital, Frederiksberg Hospital, Nordsjællands Hospital Hillerød and Aarhus Universitetshospital.

The samples will undergo plating and susceptibility testing at the Clinical Microbiological Departments of Herlev og Gentofte Hospital and Aarhus Universitetshospital.

All orthopedic departments involved are highly dedicated to this project.

Sample size calculations There are large variations in the reported frequencies of intraoperative contamination, presumably because of differences in sterile techniques and sample methods. According to the investigators' calculations a sample size of 1200 operations are needed. To demonstrate the effect of incisional drape on intraoperative contamination the investigators' have chosen to make the two groups of equal size with 600 operations in each group.

Materials and methods

The study is centered on an infection paradigm where intraoperative contamination plays a pivotal role, and the study has two main arms:

1. Intraoperative contamination (source, patient/surgeon, incisional drape).
2. Postoperative infection (correspondence with intraoperative contamination, microbiology, radiology, serology, patient-reported outcomes).

These arms together form a comprehensive study of the effects of intraoperative contamination. The study will attempt to answer all questions that arise secondary to the paradigm above, and this will be done in stages. The first stage will aim to document that patients with intraoperative contamination do indeed have a larger risk of developing post-operative infection. The first stage will also include a study of the effect of iodine impregnated incisional drape. The second stage will include highly sensitive methods of PCR and fluorescence microscopy, to demonstrate bacterial contamination and/or infection of any implants removed during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Patients of 18 years of age or older scheduled for primary knee arthroplasty surgery will be eligible for inclusion in the study

Exclusion Criteria:

* known allergy or hypersensitivity to iodine or adhesive drape
* history of infection in the knee (e.g. septic arthritis, osteomyelitis)
* active infection at another site at the time of surgery
* antibiotic use within 4 weeks before surgery
* previous enrolment in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1661 (Actual)
Dates: Start 2016-03; Primary Completion 2018-04-30 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Does Ioban prevent intraoperative microbial contamination? | approximately 2 hours. Sampling is done during surgery.
  A randomized controlled study is performed to determine the effect of iodine impregnated incisional drape on intraoperative contamination. The primary outcome is the frequency of intraoperative contamination in the projects' two arms.
Sources of intraoperative contamination | approximately 2 hours. Sampling is done during surgery.
  A prospective study is performed to assess the frequency of intraoperative contamination. During standard knee arthroplasty surgeries the samples are obtained.
  Three swabs, (Copan ESwab) will be taken during surgery. The first swab is taken from the skin of the surgical site prior to skin preparation. The second swab just after incision and will be of the wound edges.
  Intra-operative contaminants are cultured from the glove of the surgeon's dominant hand using a special glove culture technique with samples taken 30 minutes after skin incision (or before changing gloves when handling implants or using bone cement impregnated with antibiotics - whichever comes first) and the third swab is taken from the skin edges after closure of the subcutaneous tissue before closure of the skin. All the samples will be cultured and undergo susceptability testing.
  Analysis will determine the most frequent source of contamination.

SECONDARY OUTCOMES:
Postoperative infections are caused (are not caused) by intra-operative contamination. | Approximately 4 hours. Sampling done during revision surgery
  The bacteriology of postoperative, clinical infections will be compared to the intra-operative contamination.
  Kamme-Lindberg biopsies will be taken from these cases (debridements or revisions) as per usual clinical procedures. Extensive biofilm analyses will be performed of explants and biopsies and compared to extensive analyses of the glove samples from the primary procedure.
  Kamme-Lindberg biopsies will be taken from these cases (debridements or revisions) as per usual clinical procedures. Extensive biofilm analyses will be performed of explants and biopsies and compared to extensive analyses of the glove samples from the primary procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Bjarnsholt, Principal Investigator — University of Copenhagen
Locations (3):
- Denmark (3):
  - Aarhus Universitetshospital, Aarhus
  - Herlev and Gentofte Hospital, Gentofte Municipality
  - Nordsjællands Hospital, Hillerød

IPD SHARING:
Plan to Share IPD: Yes
We are making a database and keeping the records for ten years. Fellow researchers will have acces to the database.

REFERENCES:
- [Background] Jamsen E, Varonen M, Huhtala H, Lehto MU, Lumio J, Konttinen YT, Moilanen T. Incidence of prosthetic joint infections after primary knee arthroplasty. J Arthroplasty. 2010 Jan;25(1):87-92. doi: 10.1016/j.arth.2008.10.013. Epub 2008 Dec 4. PMID 19056210
- [Background] Phillips JE, Crane TP, Noy M, Elliott TS, Grimer RJ. The incidence of deep prosthetic infections in a specialist orthopaedic hospital: a 15-year prospective survey. J Bone Joint Surg Br. 2006 Jul;88(7):943-8. doi: 10.1302/0301-620X.88B7.17150. PMID 16799001
- [Background] Whitehouse JD, Friedman ND, Kirkland KB, Richardson WJ, Sexton DJ. The impact of surgical-site infections following orthopedic surgery at a community hospital and a university hospital: adverse quality of life, excess length of stay, and extra cost. Infect Control Hosp Epidemiol. 2002 Apr;23(4):183-9. doi: 10.1086/502033. PMID 12002232
- [Background] Culliford D, Maskell J, Judge A, Cooper C, Prieto-Alhambra D, Arden NK; COASt Study Group. Future projections of total hip and knee arthroplasty in the UK: results from the UK Clinical Practice Research Datalink. Osteoarthritis Cartilage. 2015 Apr;23(4):594-600. doi: 10.1016/j.joca.2014.12.022. Epub 2015 Jan 9. PMID 25579802
- [Background] Gallo J, Kolar M, Novotny R, Rihakova P, Ticha V. Pathogenesis of prosthesis-related infection. Biomed Pap Med Fac Univ Palacky Olomouc Czech Repub. 2003 Nov;147(1):27-35. doi: 10.5507/bp.2003.004. PMID 15034602
- [Background] Arnold WV, Shirtliff ME, Stoodley P. Bacterial biofilms and periprosthetic infections. J Bone Joint Surg Am. 2013 Dec 18;95(24):2223-9. doi: 10.2106/JBJS.2223. No abstract available. PMID 24498639
- [Background] Trampuz A, Zimmerli W. Prosthetic joint infections: update in diagnosis and treatment. Swiss Med Wkly. 2005 Apr 30;135(17-18):243-51. doi: 10.4414/smw.2005.10934. PMID 15965826
- [Background] Nelson CL, McLaren AC, McLaren SG, Johnson JW, Smeltzer MS. Is aseptic loosening truly aseptic? Clin Orthop Relat Res. 2005 Aug;(437):25-30. doi: 10.1097/01.blo.0000175715.68624.3d. PMID 16056022
- [Background] Lange-Asschenfeldt B, Marenbach D, Lang C, Patzelt A, Ulrich M, Maltusch A, Terhorst D, Stockfleth E, Sterry W, Lademann J. Distribution of bacteria in the epidermal layers and hair follicles of the human skin. Skin Pharmacol Physiol. 2011;24(6):305-11. doi: 10.1159/000328728. Epub 2011 Jul 15. PMID 21757977
- [Background] Al-Qahtani SM, Al-Amoudi HM, Al-Jehani S, Ashour AS, Abd-Hammad MR, Tawfik OR, Baslaim MM, Farrokhyar F. Post-appendectomy surgical site infection rate after using an antimicrobial film incise drape: a prospective study. Surg Infect (Larchmt). 2015 Apr;16(2):155-8. doi: 10.1089/sur.2013.188. Epub 2014 Aug 15. PMID 25126720
- [Background] Haliasos N, Bhatia R, Hartley J, Thompson D. Ioban drapes against shunt infections? Childs Nerv Syst. 2012 Apr;28(4):509-10. doi: 10.1007/s00381-012-1724-x. Epub 2012 Feb 22. No abstract available. PMID 22354120
- [Background] Segal CG, Anderson JJ. Preoperative skin preparation of cardiac patients. AORN J. 2002 Nov;76(5):821-8. doi: 10.1016/s0001-2092(06)61035-1. PMID 12463081
- See also: The Danish Knee Registry — http://www.sundhed.dk/sundhedsfaglig/kvalitet/kliniske-kvalitetsdatabaser/planlagt-kirugi/knaealloplastikregister/
- See also: Diagnosis and procedure codes — http://drgservice.ssi.dk/grouper/Modules/Home/